CLINICAL TRIAL: NCT03033563
Title: ICSI Outcome of Ejaculated Versus Extracted Testicular Spermatozoa in Cryptozoospermic or Severe Oligozoospermic Men
Brief Title: ICSI Outcome of Ejaculated Versus Extracted Testicular Spermatozoa
Status: Completed | Type: Observational
Sponsor: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Raef Sadek, Dr. Ahmad Raef, Adam International Hospital
Other Study IDs: 2017
Record Dates: First submitted 2017-01-21; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Intracytoplasmic Sperm Injection
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Testicular tissue versus ejaculate: Evaluation of ICSI outcome.
  Interventions: Procedure: Intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: Intracytoplasmic sperm injection — Intracytoplasmic sperm injection

SUMMARY:
The study is retrospective to compare ICSI outcome of patients with cryptozoospermia or severe oligozoospermia after use of ejaculated versus extracted testicular sperms in different cycles for the same patient.

DETAILED DESCRIPTION:
The study was carried out on couples who underwent ICSI in period 2012-2014 for male factor infertility.Patients with semen showing cryptozoospermia were candidates for inclusion in this study.

First cycle was done as ICSI with priority to ejaculated sperm; testicular sperm was used if no motile sperm was available. For failed cases a second cycle was repeated using either testicular sperm or ejaculated sperm.

Keywords:Cryptozoospermia, ejaculated spermatozoa, testicular spermatozoa, ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Couples seeking ICSI.

Exclusion Criteria:

* Couples not seeking ICSI.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile couples
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Intracytoplasmic sperm injection outcome | three years
  Pregnancy rate.

IPD SHARING:
Plan to Share IPD: No